CLINICAL TRIAL: NCT02972814
Title: Time Gain in the Diagnosis of Non-ST Elevation Myocardial Infarction by Troponin Point of Care Testing in the Emergency Room
Brief Title: Time Gain in the Diagnosis Myocardial Infarction by Troponin Point of Care Testing in the Emergency Room
Acronym: T-POCT
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Pascal Vanelderen, Prof. dr., Ziekenhuis Oost-Limburg
Other Study IDs: 16/093U
Record Dates: First submitted 2016-11-11; First posted 2016-11-23 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Non STEMI; Angina Pectoris; Angina, Stable; Angina, Unstable; Angina, Prinzmetal's
Keywords: Troponin; Point of care test; myocardial infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina Pectoris; Angina, Stable; Angina, Unstable; Angina Pectoris, Variant; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracic pain: Patients presenting to the emergency room with thoracic pain probably due to a non-STEMI
  Interventions: Device: Laboratory based troponin test; Device: Point of care based troponin test 1; Device: Point of care based troponin test 2

INTERVENTIONS:
Device: Laboratory based troponin test — acquisition of blood troponin level by Roche Cobas E 603
Device: Point of care based troponin test 1 — acquisition of blood troponin level by Radiometer EQT 90 Flex
Device: Point of care based troponin test 2 — acquisition of blood troponin level by Philips Minicare I-20

SUMMARY:
The investigators prospectively want to compare 3 clinical tests for measuring blood troponin levels in patients presenting to the emergency room with thoracic pain probably related to a myocardial infarction with regard to the time necessary to obtain the test results.

The tests are one laboratory based test and two point of care tests.

DETAILED DESCRIPTION:
Thoracic pain can be caused by a myocardial infarction. The diagnosis of a myocardial infarction can be made by an ECG (ST-elevation myocardial infarction, STEMI). However, some myocardial infarctions can also occur without ST-elevations on the ECG (non-ST-elevation myocardial infarction, non-STEMI). In the latter case, a quick acquisition of blood troponin levels is necessary to coin the diagnosis and initiate treatment. Therefore, the investigators prospectively want to compare 3 clinical tests for measuring blood troponin levels in patients presenting to the emergency room with thoracic pain probably related to a non-STEMI with regard to the time necessary to obtain the test results.

The 3 tests are:

1. A laboratory based test: Roche Cobas E 602
2. A point of care test: Radiometer AQT 90 Flex
3. A point of care test: Philips Minicare I-20

The measured timeframe is the time between venipuncture to the point the test results are known.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic pain

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency room with thoracic pain due to a non-STEMI
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
time delay until troponin test results are known | From the time of venipuncture to the time the troponin test results are known: up to 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Vanelderen, MD, PhDD, Principal Investigator — Member of Staff
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No